CLINICAL TRIAL: NCT05788354
Title: Intra-cesarean Post Placental Introducer Withdrawal IUD Insertion Technique: A New Standardized Technique for IUD Insertion During Cesarean Section. A Randomized Controlled Trial
Brief Title: Intra-cesarean Post Placental Introducer Withdrawal IUD Insertion Technique
Acronym: IUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mostafa abdel hamid seleem, professor of 0b&gyn, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: I20015
Record Dates: First submitted 2023-03-12; First posted 2023-03-28 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Intrauterine Contraceptive Device Complication

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional method (Active Comparator): IFirst, we Performed time out and verify that there were no contraindications to IUD placement:, Second, after package opening we Removed the IUD from the introducer and trimmed IUD threads to 12 cm, Third, we Grasped the IUD firmly along the stem of the device, Fourth we Stabilized the uterus using the non-dominant hand or with the aid of an assistant and advanced the IUD through the hysterotomy to the fundus, Fifth, we Removed hand and directed the IUD threads into the cervix and finally we Closed the uterine incision, took care not to incorporate the IUD strings.
  Interventions: Procedure: IUD insertion during cesarean section
- new method (Experimental): First we Performed time out and verified that there were no contraindications to IUD placement, Second, after package opening we Removed IUD from the introducer and trimmed the IUD threads to 12 cm and also trimmed the introducer to 12 cm, Third, we Loaded the IUD again inside the introducer (through the trimmed end) and kept the arms of the IUD unfolded, Forth, we removed the shoulders of the introducer, Fifth, we held the uterus and stabilized it by the non-dominant hand and guided the introducer containing the IUD strings first through the cervix then we advanced the introducer with the IUD arms unfolded to the fundus and kept the IUD their by pressing on the fundus, then we pushed the introducer gently through the cervix to the vagina, Finally, we Closed the uterine incision, took care not to incorporate the introducer or the threads and then we removed the introducer gently manually from the vagina after closure of the skin and ceiling of the wound.
  Interventions: Procedure: IUD insertion during cesarean section

INTERVENTIONS:
Procedure: IUD insertion during cesarean section — placement of IUD during cesarean section after placental delivery

SUMMARY:
This is a prospective randomized controlled study that was conducted to compare between the conventional (manual) technique of post placental IUD insertion and a new technique (intra-cesarean post placental introducer withdrawal IUD insertion technique) for IUD insertion during cesarean section regarding side effects and complications.

DETAILED DESCRIPTION:
Complete history taking and clinical examination were obtained from all cases. Lower segment cesarean section though Pfannenstiel incision was performed. Copper T380 IUDs were inserted to all participants during cesarean section after delivery of the placenta using the following techniques:

Group A (control group): (n = 420) First, the investigators Performed time out and verify that there were no contraindications to IUD placement:, Second, after package opening the investigators Removed the IUD from the introducer and trimmed IUD threads to 12 cm, Third, the investigators Grasped the IUD firmly along the stem of the device, Fourth the investigators Stabilized the uterus using the non-dominant hand or with the aid of an assistant and advanced the IUD through the hysterotomy to the fundus, Fifth, the investigators Removed hand and directed the IUD threads into the cervix and finally the investigators Closed the uterine incision, took care not to incorporate the IUD strings.

Group B (study group): (n = 420) First the investigators Performed time out and verified that there were no contraindications to IUD placement, Second, after package opening the investigators Removed IUD from the introducer and trimmed the IUD threads to 12 cm and also trimmed the introducer to 12 cm, Third, the investigators Loaded the IUD again inside the introducer (through the trimmed end) and kept the arms of the IUD unfolded, Forth, the investigators removed the shoulders of the introducer, Fifth, the investigators held the uterus and stabilized it by the non-dominant hand and guided the introducer containing the IUD strings first through the cervix then the investigators advanced the introducer with the IUD arms unfolded to the fundus and kept the IUD their by pressing on the fundus, then the investigators pushed the introducer gently through the cervix to the vagina, Finally, the investigators Closed the uterine incision, took care not to incorporate the introducer or the threads and then the investigators removed the introducer gently manually from the vagina after closure of the skin and ceiling of the wound.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women attending for elective or emergency cesarean section

Exclusion Criteria:

* upper segment cesarean scar
* cesarean for placenta previa or placenta accrete
* evident infections
* uterine anomalies
* uterine myomas
* bleeding tendency.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 788 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-04-22 (Actual)

PRIMARY OUTCOMES:
Intrauterine displacement of the IUD | 6 months
  transvaginal ultrasound : the distance from the top of the uterine cavity to the IUD which should be < 3 mm

SECONDARY OUTCOMES:
Missed or non-visualization of IUD threads | 6 months
  vaginal speculum examination: Missed or non-visualization of IUD threads by vaginal speculum examination
Discontinuation of the method | 6 months
  questionnaire
duration of surgery | 6 months
  time of surgery in minutes

CONTACTS AND LOCATIONS:
Overall Officials: mostafa AH seleem, MD, Principal Investigator — professor of ob&gyn
Locations (2):
- Egypt (2):
  - Cairo University, Cairo
  - Cairo Univesity, Cairo

IPD SHARING:
Plan to Share IPD: Yes
all the participants data collected during the study after de-identification will be available
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: beginning 1 month after publication for 5 years
Access Criteria: through direct email with the principle investigator email: mostafasaleem@kasralainy.edu.eg

REFERENCES:
- [Background] Elsokary A, Elkhyat A, Elshwaikh S. Evaluation of Post-Placental IUD Insertion during Cesarean Section at a Tertiary Care Hospital in Egypt. Open Journal of Obstetrics and Gynecology 2020;10:516-25. https://doi.org/10.4236/ojog.2020.1040046.
- [Derived] Seleem M, Sedik MM, Megahed AMM, Nabil H. Conventional manual technique of post placental IUD insertion versus intra-cesarean post placental introducer withdrawal IUD insertion technique: a new standardized technique for IUD insertion during cesarean section: a randomized controlled trial. BMC Pregnancy Childbirth. 2023 Jun 26;23(1):474. doi: 10.1186/s12884-023-05777-1. PMID 37365489